CLINICAL TRIAL: NCT03895723
Title: Minimally Invasive(Laparoscopic and Robotic) Versus Open Liver Resection for Patients With Colorectal Cancer Liver Metastases
Brief Title: Minimally Invasive Versus Open Liver Resection for Patients With Colorectal Cancer Liver Metastases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xu jianmin (Other)
Responsible Party: Sponsor-Investigator, Xu jianmin, Director of colorectal cancer center, Fudan University
Organization: Fudan University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RSRCLM-02
Record Dates: First submitted 2017-06-28; First posted 2019-03-29 (Actual); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Colorectal Liver Metastasis
Keywords: Colorectal liver metastasis; Minimally invasive surgery; Robotic surgery; Laparoscopic surgery
MeSH Terms: interventions — Laparoscopy; Conversion to Open Surgery

STUDY DESIGN:
Intervention Model Description: Arm A: minimally invasive surgery Arm B: open
Who Masked: Outcomes Assessor
Masking Description: The assessor was masking for patients treatment arms
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Minimally Invasive surgery (Experimental): the intevention of Minimally Invasive procedure contains laparoscopic and robotic liver resection
  Interventions: Procedure: laparoscopic and robotic liver resection
- Open surgery (Other): the open surgery means traditional open surgery for liver resection
  Interventions: Procedure: open surgery

INTERVENTIONS:
Procedure: laparoscopic and robotic liver resection — laparoscopic and robotic procedure for liver resection
  Arms: Minimally Invasive surgery
Procedure: open surgery — using open surgery procedure for liver resection
  Arms: Open surgery

SUMMARY:
To examine survival of patients who underwent minimally invasive versus open liver resection for colorectal cancer with liver metastases.

DETAILED DESCRIPTION:
the minimally invasive procedure contain laparoscopic or robotic surgery

ELIGIBILITY:
Inclusion Criteria:

* patients were diagnosed with colorectal cancer liver metastases
* without extra-hepatic liver metastases
* age were within 18-75 yeas
* the numbers of metastases more than 3
* the maximal tumor size of liver metastases more than 10 cm

Exclusion Criteria:

* liver metastases were unresectable.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-04-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
disease-free survival (DFS) | 3 years disease-free survival
  DFS was calculated from the date of liver resection to the date of death or recurrence or new tumors developing

SECONDARY OUTCOMES:
Overall survival (OS) | 5 years overall survival
  OS was calculated from the date of liver resection to the date of death with any reason
Sugical complications | 1 months after sugery
  According to Claivein-Dindo surgical complication system to calculate the perioperative complications related to surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Wenju Chang, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No